CLINICAL TRIAL: NCT02532972
Title: Cochlear Implantation for Treatment of Single-sided Deafness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed by IRB
Sponsor: Dr. Daniel Lee (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor-Investigator, Dr. Daniel Lee, Director, Pediatric Otology and Neurotology, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-054H
Record Dates: First submitted 2015-08-14; First posted 2015-08-26 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Total Unilateral Deafness; Unilateral Partial Deafness
MeSH Terms: interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cochlear Implant surgery (Experimental): All subjects will be part of a single arm involving placement of the Med-El MAESTRO Cochlear Implant with Flex 28 electrode array
  Interventions: Device: Med-el MAESTRO Cochlear Implant with Flex 28 electrode array

INTERVENTIONS:
Device: Med-el MAESTRO Cochlear Implant with Flex 28 electrode array — Cochlear Implant (CI) surgery followed by device activation, testing, and clinical assessment for 12 months following surgery.
  Other Names: CI; cochlear implant

SUMMARY:
This is a research study to determine whether a cochlear implantation (CI) device can improve hearing in people who are deaf in one ear (known as single-sided deafness).

DETAILED DESCRIPTION:
The goal of this study is to further investigate the role of CI in treating unilateral hearing loss and associated tinnitus. Single-sided deafness (SSD) afflicts approximately 60,000 new patients per year in the United States. The most common causes of these single-sided losses are sudden sensorineural hearing loss, Meniere's disease, trauma, and vestibular schwannoma. Patients with SSD face significant difficulty with communicating in the presence of background noise and in sound localization. Another significant problem for some SSD patients is tinnitus, which can be incapacitating and for which there are no therapies available that are considered to be of sufficient reliability to become a standard of care. Difficulty hearing in background noise and increased tinnitus can lead to significant frustration in social situations and contribute to increased isolation and a decreased quality of life. Treatment options for single sided deafness in the United States include contralateral routing of signals (CROS) hearing aids, bone-anchored hearing aids (BAHA) and use of assistive devices to improve the signal-to-noise in group situations. The first two devices take sound from the affected ear and transmit it to the unaffected ear. The last device consists of having a speaker wear a microphone and routing the signal directly to the patient's ear at a louder listening level. Although these devices can improve speech understanding in some patients, studies have shown that use of these devices does not ameliorate tinnitus or sound localization difficulties. Recent European studies have demonstrated that cochlear implantation (CI) can provide significant improvements in both perceived hearing ability and measured speech comprehension and localization in adult and pediatric patients with unilateral hearing loss. This suggests that CI may be a more effective option for this patient population than the CROS, BAHA or assistive devices.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with the ability to provide informed consent
* English as the primary language
* Medically and psychologically suitable
* Willing to receive/have received meningitis vaccinations
* Able to pay for all care received through the study, either through the subject's insurance company or through self-pay
* Able to comply with study requirements, including travel to the investigational sites
* Severe to profound sensorineural hearing loss (≥70 dB HL (decibel hearing level) thresholds between 500 and 4000 Hz) in the worse ear with ≤ 20% Consonant-Nucleus-Consonant (CNC) word scores
* Duration of single-sided deafness ≥ one year
* Tinnitus localized to the affected ear, both ears, or in the head localized to the affected ear, both ears, or in the head

  * Expected subjects include those with:
* Unilateral hearing loss secondary to viral or bacterial infection, such as meningitis or labyrinthitis
* Ménière's disease
* Sudden sensorineural hearing loss
* Vascular disease affecting the inner ear
* A combination of any number of the above conditions

Exclusion Criteria:

* Duration of single-sided deafness ≥ ten years
* Pure tone thresholds ≥ 35 dB HL at 500, 1000, 2000, and 4000 Hz in the better ear
* Consonant-Nucleus-Consonant (CNC) word scores ≤ 70% in the better ear
* Chronic otitis media in either ear
* Inner ear malformation in either ear
* Autoimmune inner ear disease (fluctuation sensorineural hearing loss in either ear)
* Evidence of retrocochlear pathology, including vestibular schwannoma
* Unilateral tinnitus in the unaffected ear
* Cochlear ossification
* Demonstrated cognitive and/or developmental challenges
* Major depression or anxiety; post-traumatic stress disorder; substance abuse
* Medical or psychological conditions that serve as contraindication to surgery
* Additional handicaps that would prevent or limit participation in evaluations
* Unrealistic patient or family expectations regarding the benefits, risks, and limitations inherent to the procedure and the prosthetic device
* Pregnant women: The investigators will specifically ask all women of childbearing age if there is a possibility they are pregnant or trying to become pregnant at the initial clinic visit; any women who are pregnant or actively trying to become pregnant will be excluded. In cases that are questionable on the day of planned surgery, a pregnancy test will be performed as per current Massachusetts Eye & Ear Infirmary anesthesia pre-operative protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Lee, MD, FACS, Principal Investigator — MEEI / MGH
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arndt S, Aschendorff A, Laszig R, Beck R, Schild C, Kroeger S, Ihorst G, Wesarg T. Comparison of pseudobinaural hearing to real binaural hearing rehabilitation after cochlear implantation in patients with unilateral deafness and tinnitus. Otol Neurotol. 2011 Jan;32(1):39-47. doi: 10.1097/MAO.0b013e3181fcf271. PMID 21068690
- [Background] Arts RA, George EL, Stokroos RJ, Vermeire K. Review: cochlear implants as a treatment of tinnitus in single-sided deafness. Curr Opin Otolaryngol Head Neck Surg. 2012 Oct;20(5):398-403. doi: 10.1097/MOO.0b013e3283577b66. PMID 22931903
- [Background] Bishop CE, Eby TL. The current status of audiologic rehabilitation for profound unilateral sensorineural hearing loss. Laryngoscope. 2010 Mar;120(3):552-6. doi: 10.1002/lary.20735. PMID 20014322
- [Background] Firszt JB, Holden LK, Reeder RM, Waltzman SB, Arndt S. Auditory abilities after cochlear implantation in adults with unilateral deafness: a pilot study. Otol Neurotol. 2012 Oct;33(8):1339-46. doi: 10.1097/MAO.0b013e318268d52d. PMID 22935813
- [Background] Kamal SM, Robinson AD, Diaz RC. Cochlear implantation in single-sided deafness for enhancement of sound localization and speech perception. Curr Opin Otolaryngol Head Neck Surg. 2012 Oct;20(5):393-7. doi: 10.1097/MOO.0b013e328357a613. PMID 22886035
- [Background] Punte AK, Vermeire K, Hofkens A, De Bodt M, De Ridder D, Van de Heyning P. Cochlear implantation as a durable tinnitus treatment in single-sided deafness. Cochlear Implants Int. 2011 May;12 Suppl 1:S26-9. doi: 10.1179/146701011X13001035752336. PMID 21756468
- [Background] Linstrom CJ, Silverman CA, Yu GP. Efficacy of the bone-anchored hearing aid for single-sided deafness. Laryngoscope. 2009 Apr;119(4):713-20. doi: 10.1002/lary.20164. PMID 19266579
- [Background] Litovsky R, Parkinson A, Arcaroli J, Sammeth C. Simultaneous bilateral cochlear implantation in adults: a multicenter clinical study. Ear Hear. 2006 Dec;27(6):714-31. doi: 10.1097/01.aud.0000246816.50820.42. PMID 17086081
- [Background] Litovsky RY, Parkinson A, Arcaroli J. Spatial hearing and speech intelligibility in bilateral cochlear implant users. Ear Hear. 2009 Aug;30(4):419-31. doi: 10.1097/AUD.0b013e3181a165be. PMID 19455039
- [Background] Saroul N, Akkari M, Pavier Y, Gilain L, Mom T. Long-term benefit and sound localization in patients with single-sided deafness rehabilitated with an osseointegrated bone-conduction device. Otol Neurotol. 2013 Jan;34(1):111-4. doi: 10.1097/MAO.0b013e31827a2020. PMID 23202156
- [Background] Niparko JK, Cox KM, Lustig LR. Comparison of the bone anchored hearing aid implantable hearing device with contralateral routing of offside signal amplification in the rehabilitation of unilateral deafness. Otol Neurotol. 2003 Jan;24(1):73-8. doi: 10.1097/00129492-200301000-00015. PMID 12544032
- [Background] Noble W, Gatehouse S. Effects of bilateral versus unilateral hearing aid fitting on abilities measured by the Speech, Spatial, and Qualities of Hearing Scale (SSQ). Int J Audiol. 2006 Mar;45(3):172-81. doi: 10.1080/14992020500376933. PMID 16579492
- [Background] Popelka GR, Derebery J, Blevins NH, Murray M, Moore BC, Sweetow RW, Wu B, Katsis M. Preliminary evaluation of a novel bone-conduction device for single-sided deafness. Otol Neurotol. 2010 Apr;31(3):492-7. doi: 10.1097/MAO.0b013e3181be6741. PMID 19816229
- [Background] Ramos A, Polo R, Masgoret E, Artiles O, Lisner I, Zaballos ML, Moreno C, Osorio A. Cochlear implant in patients with sudden unilateral sensorineural hearing loss and associated tinnitus. Acta Otorrinolaringol Esp. 2012 Jan-Feb;63(1):15-20. doi: 10.1016/j.otorri.2011.07.004. Epub 2011 Nov 30. English, Spanish. PMID 22136970
- [Background] Snapp H, Angeli S, Telischi FF, Fabry D. Postoperative validation of bone-anchored implants in the single-sided deafness population. Otol Neurotol. 2012 Apr;33(3):291-6. doi: 10.1097/MAO.0b013e3182429512. PMID 22314919
- [Background] Van de Heyning P, Vermeire K, Diebl M, Nopp P, Anderson I, De Ridder D. Incapacitating unilateral tinnitus in single-sided deafness treated by cochlear implantation. Ann Otol Rhinol Laryngol. 2008 Sep;117(9):645-52. doi: 10.1177/000348940811700903. PMID 18834065
- [Background] Vermeire K, Van de Heyning P. Binaural hearing after cochlear implantation in subjects with unilateral sensorineural deafness and tinnitus. Audiol Neurootol. 2009;14(3):163-71. doi: 10.1159/000171478. Epub 2008 Nov 13. PMID 19005250
- [Derived] Thakkar T, Knoepker J, Dennison SR, Roche JP, Litovsky RY. Spatial separation enhances speech intelligibility but increases listening effort with session-dependent variability in pupillometric measures. Front Neurosci. 2025 Nov 10;19:1655826. doi: 10.3389/fnins.2025.1655826. eCollection 2025. PMID 41333071

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cochlear Implant Surgery
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Cochlear Implant Surgery: All subjects will be part of a single arm involving placement of the Med-El MAESTRO Cochlear Implant with Flex 28 electrode array. Intervention consists of Cochlear Implant (CI) surgery followed by device activation, testing, and clinical assessment for 12 months following surgery.
Arm/Group | Cochlear Implant Surgery
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 54 [26 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Sound detection via pure-tone air conduction threshold audiometry [Mean (Full Range); unit: dB]
  Better Ear | 13.1 [6 to 24]
  Worse Ear | 96.25 [64 to 120]

OUTCOME MEASURES:

1. Primary Outcome: Sound Detection Via Pure-tone Threshold Audiometry (PTA)
Description: Sound field thresholds following cochlear implantation via pure-tone threshold audiometry. Measured in dB HL (decibels hearing level) where a lower number means more sensitive hearing and a higher number means less sensitive hearing.
Time Frame: 3, 6 and 12 months post-operatively
Population: 11 participants had surgery, but one subject opted out of additional follow-up after the 6 month visit one subject did not return for his one year followup visit following activation. As such,12 month time points only have 9 participants' data analyzed.
Measure: Mean (Full Range); unit: dB HL
Arm/Group | Cochlear Implant Surgery
Number analyzed (Participants) | 11
dB HL
  3 months post-operative: number analyzed (Participants) | 9
  3 months post-operative | 42.36 [31.25 to 47.5]
  6 months post-operative | 45.13 [33.75 to 66.25]
  12 months post-operative: number analyzed (Participants) | 9
  12 months post-operative | 39.58 [35 to 46.25]

2. Primary Outcome: Speech Perception Following Cochlear Implantation Assessed by Consonant-Nucleus-Consonant (CNC) Word Recognition Testing
Description: Ability to recognize words and sentences read by the tester from a set list at a loudness of 65 dB HL. The outcome is measured as a percent score of words recognized. The test takes place in a quiet environment.
Time Frame: Preop, 1-4 weeks, and 3, 6, and 12 months post-operatively
Population: as for outcome 1
Measure: Mean (Full Range); unit: percentage of words recognized
Arm/Group | Cochlear Implant Surgery
Number analyzed (Participants) | 11
percentage of words recognized
  Pre-operative | 4 [0 to 26]
  1-4 weeks post-surgery: number analyzed (Participants) | 10
  1-4 weeks post-surgery | 16 [0 to 34]
  3 months post-surgery: number analyzed (Participants) | 9
  3 months post-surgery | 42 [10 to 64]
  6 months post-surgery | 40 [4 to 72]
  12 months post-surgery: number analyzed (Participants) | 9
  12 months post-surgery | 46 [8 to 72]

3. Secondary Outcome: Subjective Changes in Tinnitus Following Cochlear Implantation Measured by Tinnitus Handicap Index (THI)
Description: Tinnitus severity rated by the Tinnitus Handicap Index (THI). The THI score of 0-16 means "no or slight handicap", 18 to 36 indicates "mild", 38 to 56 indicates "moderate", 58 to 76 indicates "severe", and a score of 78-100 is classified as "catastrophic handicap"
Time Frame: Preop and 12 months post-operatively
Population: 11 participants had surgery, pre and postoperative 12 month time points have 5 participants with available Tinnitus Handicap Index (THI) data 1/11 - did not have THI data available preoperatively
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Cochlear Implant Surgery
Number analyzed (Participants) | 11
score on a scale
  Pre-operative: number analyzed (Participants) | 10
  Pre-operative | 56.2 [6 to 96]
  12 months post-surgery: number analyzed (Participants) | 5
  12 months post-surgery | 6.8 [2 to 14]

ADVERSE EVENTS:
Time Frame: 1 year following surgery
Groups:
- Cochlear Implant Surgery: Med-El MAESTRO Cochlear Implant with Flex 28 electrode array
Arm/Group | Cochlear Implant Surgery
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cochlear Implant Surgery (N=11)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — hospitalization due to pneumonia
hip replacement (Musculoskeletal and connective tissue disorders) | 1 (1) — hospitalization due to hip replacement
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cochlear Implant Surgery (N=11)
dermatitis (eyelid) (Skin and subcutaneous tissue disorders) | 1 (1)
postauricular irritation (Skin and subcutaneous tissue disorders) | 1 (2)
otitis media (Ear and labyrinth disorders) | 1 (1)
incision tenderness/irritation (Skin and subcutaneous tissue disorders) | 3 (4)
tinnitus (Ear and labyrinth disorders) | 2 (2)
vertigo (Ear and labyrinth disorders) | 1 (1)
nausea and vomiting (Gastrointestinal disorders) | 1 (2)
taste disturbance (General disorders) | 3 (4)
eardrum perforation (Ear and labyrinth disorders) | 1 (1) — from IT injections
bleeding at surgical site (Blood and lymphatic system disorders) | 1 (1)
magnet retention issues requiring stronger magnet (Product Issues) | 1 (1)
oral dryness (General disorders) | 1 (1)
hyperacusis in non-implanted ear (Ear and labyrinth disorders) | 1 (1)
general otalgia and otorrhea, intermittent (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT02532972/Prot_SAP_000.pdf